CLINICAL TRIAL: NCT04398498
Title: Molecular Biomarkers in Renal Transplantation Via TruGraf® Test
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Transplant Genomics, Inc. (Industry)
Collaborators: Scripps Health (Other)
Responsible Party: Sponsor
Other Study IDs: TGRP05-US005
Record Dates: First submitted 2020-05-08; First posted 2020-05-21 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Kidney Transplant Rejection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort A: Clinical Practice: Subjects more than 60 days post-transplant
  Interventions: Diagnostic Test: Diagnostic Test: TruGraf® Testing
- Cohort B: Long Term Follow-Up: Subjects who are at least 2 years post transplant up to 5 years post-transplant
  Interventions: Diagnostic Test: Diagnostic Test: TruGraf® Testing

INTERVENTIONS:
Diagnostic Test: Diagnostic Test: TruGraf® Testing — 5 mL collection PAXgene blood sample
  Other Names: Peripheral blood gene expression profiling

SUMMARY:
The TruGraf® test is a non-invasive blood test that measures molecular gene expression profiles associated with clinical conditions previously only diagnosed by biopsy in kidney transplant recipients. The results of the TruGraf test provide additional information about the adequacy of immunosuppression and may be used to support decisions in patient management.

DETAILED DESCRIPTION:
This is a single-center, prospective, randomized study to evaluate clinical utility of TruGraf testing in patients with the following characteristics:1.Stable serum creatinine: current serum creatinine <2.3 mg/dl, <20% increase compare to the average of the previous 3 serum creatinine levels2.Kidney transplant patients who are:•more than 60 days post-transplant will be included in this study (Study A) •more than 2-yearspost-transplant but less than 5 years post-transplant (>24 months but < 60 months) will be included in this study (Study B) Scripps will enroll subjects who are post-transplant and are undergoing routine management. In Study A, patients will receive testing eight times: Month 2 (at time of surveillance biopsy) 6(at time of surveillance biopsy), 9, 12(at time of surveillance biopsy), 15, 18, 21 and 24(at time of surveillance biopsy) (plus or minus two weeks). Results of the genomic analysis will be considered in determining patient treatment plans and as a molecular guide to perform a surveillance biopsy. Clinical data elements using the Scripps EHR and cost of care will be collected for all subjects. In Study B, patients who are at least 2 years post transplant up to 5 years post-transplant will receive testing 8 times: Months 3 ,6, 9, 12, 15, 18, 21 and 24 (plus or minus two weeks)from the time of enrollment into the study. Results of the genomic analysis will be considered in determining patient treatment plans and whether any change is needed, such as whether to perform a surveillance biopsy. Clinical data elements using the Scripps EHR and cost of care will be collected for all subjects. We expect Study A to be completed 24-30months and Study B to be completed in 24-30 months.

ELIGIBILITY:
Inclusion Criteria:

* Recipient of a primary or subsequent deceased-donor or living donor kidney transplantation.
* Stable serum creatinine (current serum creatinine <2.3 mg/dl, <20% increase compared to the average of the previous 3 serum creatinine levels).
* Kidney transplant patients who are: > 60 days post-transplant (Cohort A); > 2-years post-transplant (Cohort B)

Exclusion Criteria:

* Need for combined organ transplantation with an extra-renal organ and/or islet cell transplant.
* Recipients of previous non-renal solid organ and/or islet cell transplantation.
* Infection with HIV.
* Infection with BK.
* Patients that have nephritic proteinuria (urine protein >3 gm/day).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Kidney transplant recipients
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-04-13 (Actual); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
Cohort A: Percent or total number of patients who physicians decided could forego a surveillance biopsy due to TruGraf results | 12 months post-transplant
Cohort A: Percent or total number of patients who physicians decided could forego a surveillance biopsy due to TruGraf results | 24 months post-transplant
Cohort A: Correlation of TruGraf test results with surveillance biopsy | 2 years
Cohort A and B: Banff pathology | 2 years
  Banff pathology will be assessed and compared to TruGraf results.
Cohort A and B: Renal graft function | 2 years
  Renal graft function will be assessed by measuring Estimated Glomerular Filtration Rate (eGFR).
Cohort A and B: Renal graft function | 2 years
  Renal graft function will be assessed by measuring serum creatinine (sCr) levels.
Cohort A and B: Cost of patient care | 2 years
  The cost of patient care will be evaluated by measuring the total health care spending for health care services provided during the study period.

SECONDARY OUTCOMES:
Incidence of death | 2 years
Incidence of graft loss | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Patty West-Thielke, PharmD, Study Director — Transplant Genomics, Inc.
Locations (1):
- Scripps Clinic, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rana A, Gruessner A, Agopian VG, Khalpey Z, Riaz IB, Kaplan B, Halazun KJ, Busuttil RW, Gruessner RW. Survival benefit of solid-organ transplant in the United States. JAMA Surg. 2015 Mar 1;150(3):252-9. doi: 10.1001/jamasurg.2014.2038. PMID 25629390
- [Background] Matas AJ, Gillingham KJ, Humar A, Kandaswamy R, Sutherland DE, Payne WD, Dunn TB, Najarian JS. 2202 kidney transplant recipients with 10 years of graft function: what happens next? Am J Transplant. 2008 Nov;8(11):2410-9. doi: 10.1111/j.1600-6143.2008.02414.x. PMID 18925907
- [Background] Lamb KE, Lodhi S, Meier-Kriesche HU. Long-term renal allograft survival in the United States: a critical reappraisal. Am J Transplant. 2011 Mar;11(3):450-62. doi: 10.1111/j.1600-6143.2010.03283.x. Epub 2010 Oct 25. PMID 20973913
- [Background] Montgomery RA. One kidney for life. Am J Transplant. 2014 Jul;14(7):1473-4. doi: 10.1111/ajt.12772. Epub 2014 May 9. No abstract available. PMID 24816339
- [Background] Matas AJ, Smith JM, Skeans MA, Thompson B, Gustafson SK, Stewart DE, Cherikh WS, Wainright JL, Boyle G, Snyder JJ, Israni AK, Kasiske BL. OPTN/SRTR 2013 Annual Data Report: kidney. Am J Transplant. 2015 Jan;15 Suppl 2:1-34. doi: 10.1111/ajt.13195. PMID 25626344
- [Background] Waldmann H. Drug minimization in transplantation: an opinion. Curr Opin Organ Transplant. 2014 Aug;19(4):331-3. doi: 10.1097/MOT.0000000000000099. No abstract available. PMID 24991978
- [Background] Racusen LC, Solez K, Colvin RB, Bonsib SM, Castro MC, Cavallo T, Croker BP, Demetris AJ, Drachenberg CB, Fogo AB, Furness P, Gaber LW, Gibson IW, Glotz D, Goldberg JC, Grande J, Halloran PF, Hansen HE, Hartley B, Hayry PJ, Hill CM, Hoffman EO, Hunsicker LG, Lindblad AS, Yamaguchi Y, et al. The Banff 97 working classification of renal allograft pathology. Kidney Int. 1999 Feb;55(2):713-23. doi: 10.1046/j.1523-1755.1999.00299.x. PMID 9987096
- [Background] Rush D, Nickerson P, Gough J, McKenna R, Grimm P, Cheang M, Trpkov K, Solez K, Jeffery J. Beneficial effects of treatment of early subclinical rejection: a randomized study. J Am Soc Nephrol. 1998 Nov;9(11):2129-34. doi: 10.1681/ASN.V9112129. PMID 9808101
- [Background] Nankivell BJ, Chapman JR. The significance of subclinical rejection and the value of protocol biopsies. Am J Transplant. 2006 Sep;6(9):2006-12. doi: 10.1111/j.1600-6143.2006.01436.x. Epub 2006 Jun 22. PMID 16796717
- [Background] Legendre C, Thervet E, Skhiri H, Mamzer-Bruneel MF, Cantarovich F, Noel LH, Kreis H. Histologic features of chronic allograft nephropathy revealed by protocol biopsies in kidney transplant recipients. Transplantation. 1998 Jun 15;65(11):1506-9. doi: 10.1097/00007890-199806150-00020. PMID 9645814
- [Background] Seron D, Moreso F. Protocol biopsies in renal transplantation: prognostic value of structural monitoring. Kidney Int. 2007 Sep;72(6):690-7. doi: 10.1038/sj.ki.5002396. Epub 2007 Jun 27. PMID 17597702
- [Background] Heilman RL, Devarapalli Y, Chakkera HA, Mekeel KL, Moss AA, Mulligan DC, Mazur MJ, Hamawi K, Williams JW, Reddy KS. Impact of subclinical inflammation on the development of interstitial fibrosis and tubular atrophy in kidney transplant recipients. Am J Transplant. 2010 Mar;10(3):563-70. doi: 10.1111/j.1600-6143.2009.02966.x. Epub 2010 Feb 1. PMID 20121731
- [Background] Rush DN, Henry SF, Jeffery JR, Schroeder TJ, Gough J. Histological findings in early routine biopsies of stable renal allograft recipients. Transplantation. 1994 Jan;57(2):208-11. doi: 10.1097/00007890-199401001-00009. PMID 8310509
- [Background] Kirk AD, Jacobson LM, Heisey DM, Radke NF, Pirsch JD, Sollinger HW. Clinically stable human renal allografts contain histological and RNA-based findings that correlate with deteriorating graft function. Transplantation. 1999 Nov 27;68(10):1578-82. doi: 10.1097/00007890-199911270-00024. PMID 10589958
- [Background] Moreso F, Ibernon M, Goma M, Carrera M, Fulladosa X, Hueso M, Gil-Vernet S, Cruzado JM, Torras J, Grinyo JM, Seron D. Subclinical rejection associated with chronic allograft nephropathy in protocol biopsies as a risk factor for late graft loss. Am J Transplant. 2006 Apr;6(4):747-52. doi: 10.1111/j.1600-6143.2005.01230.x. PMID 16539631